CLINICAL TRIAL: NCT04924738
Title: A Prospective Observational Trial of Factors Involved in the Intergenerational Transmission of the Non-communicable Disorders - Female Obesity Cohort and Intervention Study Group.
Brief Title: Female Obesity Cohort and Intervention Study Group (MOCART Study Group)
Acronym: MOCART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pawel Bogdanski, Director of the Department of Treatment of Obesity, Metabolic Disorders and Clinical Dietetics, Poznan University of Medical Sciences
Other Study IDs: 102/19; 525/17 (Other: Poznan University of Medical Sciences - Bioethics Board)
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Endocrine; Pregnancy in Diabetic; Child Obesity; Hypertension in Pregnancy
Keywords: DOHaD - developmental origins of health and disease; hyperglycemia in pregnancy; gestational weight gain; adipokines; endothelium dysfunction; large for gestational age; macrosomia; early life origins of health and disease
MeSH Terms: conditions — Obesity; Pregnancy in Diabetics; Pediatric Obesity; Hypertension, Pregnancy-Induced; Disease; Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, serum, hair, cord blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MOZART_SG: Women treated for hyperglycemia in pregnancy. Observational data are to be collected at follow-up visits during pregnancy, at delivery and postpartum.
  Interventions: Behavioral: Monitoring and lifestyle

INTERVENTIONS:
Behavioral: Monitoring and lifestyle — Dietary and lifestyle modification recommended for pregnant women with hyperglycemia detected in pregnancy.

SUMMARY:
This prospective observational trial includes women with high risk pregnancies complicated with hyperglycemia in pregnancy and excessive body weight. The participants are enrolled when pregnant and monitored throughout pregnancy and delivery until the offspring is 6 months old. This research addresses the question which risk factors for non-communicable disorders such as hypertension, obesity, type 2 diabetes for a woman and her offspring can be detected during pregnancy and in early childhood.

DETAILED DESCRIPTION:
The available epidemiological data clearly indicate a significant increase in the percentage of people with obesity and the metabolic syndrome in the population of women of reproductive age. These diseases predispose to the onset of type 2 diabetes at a young age and accelerate the risk of cardiovascular diseases, while in pregnant population they constitute a serious risk factor for gestational diabetes.

Recent decades have brought a growing amount of evidence from prospective studies indicating the adverse impact of gestational diabetes on the health prognosis of the mother and her child. In the short-term perspective, hyperglycemia in pregnancy constitutes a risk factor for numerous maternal-fetal complications, in particular hypertensive diseases in pregnancy, excessive fetal growth, intrapartum complications induced by excessive birth weight of the newborn, which can result in intrapartum neonatal asphyxia or maternal postpartum haemorrhage. Gestational diabetes is also associated with an increased risk of fetal intrauterine death in late pregnancy, during delivery or postpartum.

However, there is growing evidence of the adverse effects of gestational diabetes on long-term health outcomes of the mother and her offspring, even when glucose tolerance disorders are resolved after delivery. Hyperglycemia detected in pregnancy is a strong risk factor for the development of type 2 diabetes within several years after experiencing a complicated pregnancy. Moreover, maternal hyperglycemia has been shown to adversely affect the long-term risk of obesity, metabolic syndrome, pre-diabetes, and type 2 diabetes in the offspring of this pregnant population. This relationship is so clear that it is the exposure of the fetus to the abnormal intrauterine metabolic environment that is considered to be one of the leading causes of the significantly increased prevalence of the aforementioned civilization diseases among children and adolescents.

The authors of the study expect that the obtained results will provide important data enabling early identification of the population that can benefit most measurably from the diagnosis and possible treatment of conditions predisposing to the non-communicable diseases. The authors believe, that this study will identify specific maternal characteristics that could be targets for individualized interventions modifying risk factors of civilization diseases in mothers and their offspring. The authors expect that the measurable effect of the research will be achievable in the short term - in the form of reduction of maternal-fetal complications characteristic of pregnancy complicated with obesity and / or gestational diabetes (maternal "diabesity"), and in the long term - in the form of improvement of the incidence rates of non-communicable disorders in the population of pregnant women of a risk profile similar to this presented by the cohort included in the study.

Research objectives:

* identification of epigenetic risk factors of intergenerational glucose tolerance disorders and examining the possibility of their modification so as to break the intergenerational "vicious circle" of metabolic syndrome and lifestyle diseases resulting from it;
* identification of mechanisms responsible for the intergenerational transmission of classic and "new" risk factors of non-communicable diseases;
* gather information for future trials on development and evaluation of interventions aimed at reducing the effects of the intergenerational "vicious circle" of obesity, insulin resistance and diseases related to lifestyle.

The protocol includes the following visits:

V0 - recruitment, V1 - gestational age 28-32 weeks, V2 - gestational age 36-38 weeks, V3 - delivery, V4 - six weeks postpartum, V5 - six months postpartum

At the V0, the researchers will collect detailed information concerning demographics, anthropometrics, past diseases, pregnancy-related conditions, lifestyle and dietary habits

At the V1, V2, V4 and V5, the researchers collect data regarding maternal glucose levels and body weight, perform noninvasive tests of cardiovascular function and collect biological material to be aliquoted, frozen and stored for further examination of biomarkers of oxidative stress, fat tissue function, inflammation, insulin resistance, clotting system, cardiometabolic risk; also information regarding fetal growth (V1,V2) and child's anthropometrics and development (V4, V5) will be collected.

At the V3, the researchers collect a detailed information regarding delivery and neonatal anthropometrics, and collect samples of placenta and cord blood to be aliquoted, frozen and stored for further examination (see above).

At the V6, the researchers collect information regarding maternal dietary and lifestyle habits, perform noninvasive tests of cardiovascular function and collect biological material to be aliquoted, frozen and stored for further examination of biomarkers of oxidative stress, fat tissue function, inflammation, insulin resistance, clotting system, cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* a woman in a singleton pregnancy referred to the Department of Reproduction, Poznan University of Medical Sciences
* maternal BMI (body mass index): 27 kg/m2 or above
* hyperglycemia detected in pregnancy according to the Polish Diabetes Association criteria, 2017
* delivery in the University Hospital

Exclusion Criteria:

* fetal malformation
* any serious maternal conditions that might hamper patient's participation in the tiral

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Tertiary level of perinatal care unit.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-12-03 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
maternal weight before delivery | measured at term, within a week before delivery
  kg
maternal weight in the early pregnancy | measured after a viable pregnancy confirmed until a gestational age of 12 weeks
  kg
birth weight | neonate's weight measured immediately after birth
  g

SECONDARY OUTCOMES:
maternal blood pressure at the term | measured at term, within a week before delivery
  mmHg
average maternal fasting glucose at the term | measured seven times within two weeks before delivery
  mg/dl
average maternal postprandial glucose at the term | measured one hour after main meals, twenty-one times within two weeks before delivery
  mg/dl
maternal HbA1c at the term | glycated haemoglobin measured within a month before delivery
  percent [%]

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Wender-Ożegowska, prof., Study Director — Head of the Department of Reproduction
Locations (1):
- Department of Reproduction, Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided